CLINICAL TRIAL: NCT01236651
Title: Comparison Between Meperidine and Drotaverine Regarding the Effect on the Duration of the First Stage of Labor in Full Term Primigravidae
Brief Title: Meperidine Versus Drotaverine Regarding the Effect on the Duration of the First Stage of Labor in Full Term Primigravidae
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: ain shams university, ain shams university
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: dr hegab protocol
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Effect of Meperidine or Drotaverine on Effacement and Dilatation of the Cervix During Labor in Full Term Primigravidae
MeSH Terms: interventions — Meperidine; drotaverin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- meperidine and duration of 1st stage of labor (Experimental): meperidine 100mg i.v in 1st stage of labor and calculate the duration of the 1st stage of labor
  Interventions: Drug: Meperidine
- drotaverine and duration of 1st stage of labor (Experimental): drotaverine 40mg i.v in 1st stage of labor and calculate the duration of the 1st stage of labor
  Interventions: Drug: Drotaverine

INTERVENTIONS:
Drug: Meperidine — administer 100mg meperidine i.v during the 1st stage of labor and calculate the duration of this stage of labor
  Arms: meperidine and duration of 1st stage of labor
Drug: Drotaverine — administer 40mg drotaverine i.v during the 1st stage of labor and calculate the duration of this stage of labor
  Arms: drotaverine and duration of 1st stage of labor

SUMMARY:
Comparison Between Meperidine and Drotaverine Regarding the Effect on the Duration of the First Stage of Labor in Full Term Primigravidae

DETAILED DESCRIPTION:
Comparison Between Meperidine and Drotaverine Regarding the Effect on the Duration of the First Stage of Labor in Full Term Primigravidae

Protocol of Thesis Submitted for partial fulfillment of master degree in Obstetrics & Gynecology

The aim of this work is to compare and to evaluate the efficacy of drotaverine hydrochloride versus meperidine hydrochloride on the duration of the 1st stage of labor.

ELIGIBILITY:
Inclusion Criteria: ● primigravida.

* Singleton pregnancy.
* Term gestation i.e, 38-41 weeks.
* Sure, reliable dates documented by ultrasound in the 1st half of pregnancy.
* Vertex presentation with occipito anterior position.
* Efficient uterine contractions at a rate of at least 3 to 4 contractions every 10 minutes, each contraction lasting for at least 40 seconds.

Exclusion Criteria: ● Abnormal presentation or occipito posterior position.

* Multiple pregnancies.
* Cephalo-pelvic disproportion.
* Cervical surgery in the past or history of cervical injury.
* Patients on antihypertensive therapy.
* Known hypersensitivity to drotaverine or meperidine.
* If any other spasmolytic agent had been used within 48 hours.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-04 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
the duration of the first stage of labor | 6 monthes
  the primary outcome is to evaluate whether meperidine or drotaverine is more effective in shortening the duration of the 1st stage of labor
effect on the duration of the 1st stage of labor | 6 monthes
  the primary outcome is to evaluate whether meperidine or drotaverine is more effective on the duration of the 1st stage of labor

SECONDARY OUTCOMES:
effect on pain | 6 monthes

CONTACTS AND LOCATIONS:
Locations (1):
- Mahmoud, Cairo, Egypt